CLINICAL TRIAL: NCT05189834
Title: Effects of GELSECTAN® Administration on Covert Hepatic Encephalopathy (CHE) in Patients With Cirrhosis.
Brief Title: GELSECTAN® and Covert Hepatic Encephalopathy
Acronym: GELSECTAN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was not performed because logistical problems
Sponsor: Consorci Sanitari de l'Alt Penedès i Garraf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSAPG-3
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Covert Hepatic Encephalopathy
Keywords: Covert Hepatic Encephalopathy; Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment sequence A (Other): Patients will follow the following treatment sequence:
  1. Treatment with Gelsectan® (30 days)
  2. Washout period (15 days)
  3. Treatment with placebo (30 days)
  Interventions: Dietary Supplement: Gelsectan
- Treatment sequence B (Other): Patients will follow the following treatment sequence:
  1. Treatment with placebo (30 days)
  2. Washout period (15 days)
  3. Treatment with Gelsectan® (30 days)
  Interventions: Dietary Supplement: Gelsectan

INTERVENTIONS:
Dietary Supplement: Gelsectan — Xyloglucan, vegetable protein and xylooligosaccharides

SUMMARY:
Randomized crossover pilot clinical trial in which 10 cirrhotic patients with covert hepatic encephalopathy (CHE) will be assigned to take GELSECTAN® (TID) or placebo for 30 days. After a washout period of 15 days, the treatment branches will be interchanged.

The objective of the trial is to obtain pilot variances to design a phase II trial, in which the efficacy of the treatment will be tested. As an exploratory objective, the efficacy of the product in the treatment of covert hepatic encephalopathy will be analyzed.

Main endpoint Improvement in CHE after 30 days of treatment with GELSECTAN®, measured by the Psychometric hepatic encephalopathy score (PHES)

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85 years.
2. Liver cirrhosis defined by a previous liver biopsy or by clinical data.
3. Presence of minimal hepatic encephalopathy (MHE) defined by two psychometric methods (PHES and / or S-ANT and / or Sloop-test).
4. Adequately informed patients who grant their written consent to participate in the study.

Exclusion Criteria:

1. Alternative neurological diagnosis.
2. Hepatic encephalopathy stage ≥2 using the adapted West-Haven scale.
3. Terminal disease. At the discretion of the doctor, where the patient is in an irreversible situation, in which hepatic encephalopathy is a final manifestation.
4. Presence of Acute-on-chronic liver failure defined by the presence of decompensated liver cirrhosis with severe organ or multi-organ failure.
5. MELD score greater than 25 at the time of inclusion.
6. Hospitalization for any reason.
7. Neurological or psychiatric comorbidity that makes the evaluation of hepatic encephalopathy difficult. This includes patients with mental illnesses (dementia, cerebrovascular disease with sequelae, Parkinson's disease, schizophrenia).
8. Active digestive bleeding. Before inclusion, there must have been a 48-hour period without signs of bleeding.
9. Patients with hypersensitivity or allergy to any of the components of GELSECTAN® (grape, pea).
10. Clinical situations in which the administration of oral feeding is contraindicated.
11. Active oncological processes, including hepatocarcinoma.
12. Active infection of any origin.
13. Acute renal failure (AKI). Defined by the current diagnostic criteria of the KDIGO group (Kidney Disease Improving Global Outcomes).
14. Dehydration Diagnosed by physical examination of the patient.
15. Severe hyponatremia. Defined by plasma sodium <130 mEq / dl.
16. Concomitant use of sedative drugs, such as benzodiazepines, morphic or derivatives (methadone, tramadol ...)
17. Active drug and/or alcohol use. In each case of clinical suspicion of drug use, an analysis of toxins in urine will be carried out, which includes cocaine, cannabis, opiates. All patients with confirmed alcohol consumption greater than 3 UBD in men or 2 UBD in women will be excluded.
18. Consumption of drugs currently indicated for the treatment of HE: Lactulose, lactitol and antibiotics.
19. Participation in another clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-11 (Estimated); Primary Completion 2022-05-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Covert Hepatic Encephalopathy change | 30 days
  Covert Hepatic Encephalopathy change after 30 days of treatment with GELSECTAN®, by means of the Psychometric hepatic encephalopathy score (PHES), being patients classified as having MHE when their PHES is less than -4

CONTACTS AND LOCATIONS:
Locations (1):
- Consorci Sanitari Alt'Pènedes i Garraf, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF